CLINICAL TRIAL: NCT02356848
Title: STEP UP to Avert Amputation in Diabetes
Acronym: STEP UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E1858-R
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Diabetes; Foot Ulcer
Keywords: self-care; self-monitoring; secondary prevention; foot ulcer; Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tailored intervention (TI) (Experimental): Participants in this arm will receive a comprehensive intervention based on the Transtheoretical Model and Prospect Theory with the counseling being delivered by health counselors using MI principles. This arm will have biweekly calls for the first two months and then monthly calls for the next four months followed by texts or mailings for months 7-18 with the frequency determine by level of treatment adherence.
  Interventions: Behavioral: Tailored Intervention (TI)
- Current Practice (CP) (Placebo Comparator): This group will receive all the enhancements that the VA has targeted to improve foot risk in diabetes including full EMR functionality, clinical reminders to improve care, and Patient-Centered Medical Home (PCMH) implementation with its benefits for diabetes care. To control for attention and preserve blinding, this group will receive calls and mailings focusing on providing education and prevention strategies for health conditions such as colorectal cancer, influenza, insomnia, vision, dementia, and oral disease. This arm will have biweekly calls for the first two months and then monthly calls for the next four months followed by texts or mailings for months 7-18 with the frequency determine by level of treatment adherence to general health recommendations
  Interventions: Behavioral: Current Practice (CP)

INTERVENTIONS:
Behavioral: Tailored Intervention (TI) — Participants in this arm will receive a comprehensive intervention based on the Transtheoretical Model and Prospect Theory with the counseling being delivered by health counselors using MI principles.
  Arms: Tailored intervention (TI)
Behavioral: Current Practice (CP) — this group will receive calls and mailings focusing on providing education and prevention strategies for health conditions such as colorectal cancer, influenza, insomnia, vision, dementia, and oral disease.
  Arms: Current Practice (CP)

SUMMARY:
This study will evaluate a comprehensive tailored behavioral intervention aimed to improve foot self-care and self-monitoring (combined with dermal thermometry) to prevent recurrent ulcers in Veterans at highest risk of amputation. This intervention may be a novel strategy for improving self-care and early detection of foot abnormalities in this at-risk population using psychological theories to target multiple health behaviors simultaneously. This could be an efficient and cost-effective approach to improve diabetes-related foot health behavior, and other risk factors in patients who are vulnerable to devastating consequences related to amputation.

DETAILED DESCRIPTION:
Veterans with diabetes who have had a previous ulcer are at highest risk for new ulcers and amputation, particularly if they have neuropathy or vascular disease and have poor foot self-care or nonadherence to diet, medication, and exercise recommendations. It is difficult to activate at-risk patients to improve self-care and detect foot abnormalities or inflammation at an early stage.

Proposed is a randomized controlled trial testing the effectiveness of a comprehensive tailored intervention (TI) aimed to improve self-care and self-monitoring (including dermal thermometry) through behavioral counseling. The primary specific aim is to evaluate if TI reduces the proportion of recurrent ulcers at 18 months compared to the current practice (CP) group. The secondary specific aims are to evaluate the impact of TI on time to ulceration, quality of life (QOL), plantar pressure, physical activity and foot care skills compared to the CP group.

The investigators will recruit adults with diabetes who have had a previously healed ulcer. The intervention will be standardized and fidelity of the intervention will be maintained. Using a blinded randomized controlled trial (RCT), the investigators will test the effect of TI in relation to CP. Key outcomes are ulceration, quality of life (QOL), plantar pressure, physical activity and foot care skills. Outcomes will be measured at baseline, 6, 12 and 18 months. All analyses will be intent-to-treat.

This study will evaluate a comprehensive tailored intervention targeting multiple behaviors related to self-care and amputation risk. This study applies advanced behavioral theories to intervene to improve care for veterans at risk for amputation combined with dermal thermometry. If this promising theory-driven approach can work in a clinical setting where improvements in foot care are urgently needed for these vulnerable Veterans with a previous ulcer, it will be an important scientific contribution that could lower the risk of recurrent ulcers and amputation in Veterans with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (21 years) with Type 2 diabetes
* History of healed diabetic foot ulcer (>3 months)
* Diabetes therapy for > 6 months
* An available phone and receiving continuity of care at the VA (at least 2 primary care visits in the previous 1.5 years at the recruitment site)

Exclusion Criteria:

* Patients with an active foot ulcer
* Acute cardiovascular disease (CVD) events < 3 months ago
* Poor estimated short-term survival (< 1 year)
* Recent major surgery (< 3 months)
* Prior foot amputation
* Inability to exercise
* Temporary residence in the area
* Inability to provide consent will be excluded

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2015-09-03 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Ulceration | 18 months
  High-resolution standard view digital photographs of the feet and footwear will be obtained and reviewed by the investigators blinded to group assignment, and a suspected ulcer or nonulcerative plantar lesion below the malleoli will be referred to a panel of three blinded (as to group assignment) adjudicators, all clinical experts. Lesions will be judged as absent/nonulcerative lesion/ulcer; involving/not involving the plantar surface (defined as involving the weight-bearing surface of the foot); and related to metatarsal head (MTH)/not related to MTH. Adjudicators will not confer with each other or with the study staff, and the majority opinion will be taken as the final judgment. Ulcers will be judged to be present if the integrity of both the epidermis and dermis is broken. When ulcers occur in between study visits, the adjudication committee will review the medical records and make the determination.

SECONDARY OUTCOMES:
Foot care skills | 18 months
  The investigators will use the Veterans foot self-care education and behavior survey to assess different subscales of foot care. The investigators will measure basic foot-care education, extended foot-care education, basic professional foot care, extended professional foot care, basic foot self-care, and extended foot self-care using this survey that was developed and validated in high-risk Veterans.
General Quality of Life | 18 months
  The SF-36 will assess general well-being, and physical and mental health
Foot health-specific quality of life | 18 months
  The Foot Health Status Questionnaire (FHSQ),93 a reliable and valid instrument, will measure foot health-related quality of life.
plantar pressure | 18 months
  Plantar pressure measurements will be used to identify specific areas of high pressure under the foot. Plantar forces and pressures will be recorded during level barefoot walking using the TekScan High Resolution (HR) MatScan system.
step count | 18 months
  Step count will be assessed via accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Sundar Natarajan, MD MSc, Principal Investigator — Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY
Locations (1):
- Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No